CLINICAL TRIAL: NCT05521061
Title: The Effects of Synthetic Human Milk Oligosaccharides on Gut Microbiota, Pancreas Beta Cell Preservation and Metabolic Control in Children With Type 1 Diabetes Mellitus
Brief Title: The Effect of Human Milk Oligosaccharides in Children With Type 1 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Acibadem University (Other); Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Raika Durusoy, Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 121S556
Record Dates: First submitted 2022-05-15; First posted 2022-08-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Type1diabetes
Keywords: Diabetes mellitus; intestinal microbiota; oligosaccharides; human milk
MeSH Terms: conditions — Diabetes Mellitus | interventions — 2'-fucosyllactose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.5 g/day 2-fucosyllactose (Experimental): 1.5 g/day of human milk oligosaccharides will be supplemented in the first intervention group.
  Interventions: Dietary Supplement: 2-fucosyllactose
- 3 g/day 2-fucosyllactose (Experimental): 3 g/day of human milk oligosaccharides will be supplemented in the second intervention group.
  Interventions: Dietary Supplement: 2-fucosyllactose
- Maltodextrine (Placebo Comparator): The placebo group will receive maltodextrin as a placebo at a dose with no effect on metabolic control.
  Interventions: Dietary Supplement: 2-fucosyllactose

INTERVENTIONS:
Dietary Supplement: 2-fucosyllactose — Volunteers will be visited to provide the investigational product/placebo to the diets of the patients included in the study for 3 months, and the use of the investigational product/placebo will be monitored. Parents will be trained by their fellows to provide synthetic breast milk oligosaccharides/placebo, the products to be used in the study will be provided by the scholars on a weekly basis, and their daily intake and possible problems will be monitored through weekly interviews. In this study, it is planned to supplement the diet of the placebo group with 1.5 g/day maltodextrins to approximately half of the diet and to supplement the other half with 3 g/day maltodextrins, after the group was randomized within itself. Effects of these doses on metabolic control are not expected. Maltodextrine is in powder form, its dosage of up to 3 g/day has a negligible effect on blood glucose, it has a neutral taste, it is cheap and easy to find, and it is safe and ineffective.

SUMMARY:
Type 1 diabetes mellitus (DM) is an autoimmune disease characterized by absolute insulin deficiency, defined as insulin-dependent diabetes mellitus and develops due to autoimmune damage of beta cells in the pancreas. Approximately 425 million people worldwide are diabetic patients, 5% to 10% of whom are T1DM. In the majority of type 1 DM prevention studies, the main aim is to stop beta cell destruction. Primary prevention studies aim to prevent or alter exposure to environmental stimuli before autoimmunity is developed. Secondary prevention studies address interventions in the autoimmune processes that cause betacell destruction. Tertiary prevention studies include interventions to stop or reverse beta-cell destruction after clinical diagnosis of type 1 DM. Despite all technological advances, type1DM has not shown a permanent improvement in metabolic control over the last 5 years. Breast milk provides protection against Type 1 DM through the prevention of diabetogenic infections, delaying exposure to diet antigens including cow's milk, and the ability to produce healthy intestinal microbiota. Xiao et al. (2018) published in Nature, investigated the effect of human milk oligosaccharides on non-obese diabetic rats, where it was found that it improved intestinal flora and insulitis scores and brought the blood glucose level closer to the optimum level.

This study is expected to fill the gap in the literature about dose-dependent efficacy and placebo of breastmilk oligosaccharides in diabetic humans. This project will investigate 1) the possible contribution of 2-FL oligosaccharides to the disease's metabolic control 2) their effects on beta-cell preservation in the pancreas 3)their effects on intestinal microbiota 4) whether there is a doseresponse relationship as compared to placebo among type 1 diabetic children. This project is designed as a double-blind randomized placebo-controlled experiment lasting for 36 months. The proposed research population consists of 111 children aged 4-16-year-old who were diagnosed with Type 1 DM at the Department of Pediatric Endocrinology of Ege University. The sample size was calculated as 111 with an effect size of 0.33, an error of 0.05 and a power of 80% using the F-test group (for a numerical variable such as blood glucose) for 3 groups. It is planned that the two intervention arms consist of 37 volunteers and the placebo group of 37 volunteers. In the research, 1.5 g/day of human milk oligosaccharides will be supplemented in the first intervention group and 3 g/day for the second intervention group. The placebo group will receive maltodextrin as a placebo at a dose with no effect on metabolic control. Patients included in the study will be provided human milk oligosaccharides for 3 months and will be under follow-up for 12 months. All variables, mainly C-peptide, HbA1c, immunoglobulins, lymphocytes and faecal analysis will be examined. The project aims to ameliorate the microbiota profile, optimize C-peptide levels, reduce exogenous insulin dependence through the provision of 2-FL from human milk oligosaccharides and develop a more applicable, acceptable and an innovative method in the metabolic control of the disease. It is believed that the psychosocial and economic burdens of the disease will be reduced by increasing the metabolic control of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 48 months of age
* Diagnosis period <100 days, in the early stage
* Exogenous insulin requirement > 0.5 U/kg/day in the late-stage
* Positive at least one autoantibody associated with type 1 DM (ICA, IAA, GADA)
* C-peptide level <0.2 nmol/L during MMTT
* Between the 3rd percentile and the 97th percentile weight for age (between -2SD and +2SD)

Exclusion Criteria:

* Being breastfed despite the age of 48 months
* Failure to meet the diagnostic criteria for autoimmune type 1 DM (autoantibody negative)
* Co-morbidity illness
* To have taken antibiotics, probiotics, prebiotics and inflammatory drugs in the last one month before participating in the study or during the study

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
C peptide level | 12 weeks
HbA1C levels | 12 weeks

SECONDARY OUTCOMES:
Pancreas autoantibody levels | 12 weeks
Total daily dose of insulin | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No